CLINICAL TRIAL: NCT04533542
Title: Nicotine Vapor Specific Sensory Measurement
Status: Completed | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: I 471719; NCI-2019-06972 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 471719 (Other: Roswell Park Cancer Institute); U54CA238110 (Other Grant/Funding Number: National Institute of Health)
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Substance-Related Disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Arm I (3 video or telephone conferences): Participants attend up to 3 video or telephone conferences over 2 hours each with a minimum of 24 hours and maximum of 1 week between sessions. Participants take a fixed number of puffs on 3 randomly assigned conditions (combinations of carrier and nicotine concentrations).
  Interventions: Other: Measurement; Other: Questionnaire Administration
- Arm II (2 video or telephone conferences): Participants attend up to 2 video or telephone conferences over 2 hours each with a minimum of 24 hours and maximum of 1 week between sessions. Participants take a fixed number of puffs on a nicotine-free condition and 3 randomly assigned conditions (combinations of carrier concentration and nicotine form).
  Interventions: Other: Measurement; Other: Questionnaire Administration

INTERVENTIONS:
Other: Measurement — Undergo sensory measurements
  Other Names: Measure; {Measure}
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial aims to develop reliable and valid measures of sensory experiences unique to e-cigarette use. Regardless of whether flavorings show evidence of toxicity in a biological sense, they may nonetheless increase harm by other means, such as increasing appeal, decreasing risk perceptions, or masking harshness or irritation that might lead users to discontinue use.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Study that flavors might be related to the phenomenon of 'indirect' toxicity.

OUTLINE: Participants are randomized to 1 of 2 conditions.

CONDITION I: Participants attend up to 3 video or telephone conferences over 2 hours each with a minimum of 24 hours and maximum of 1 week between sessions. Participants take a fixed number of puffs on 3 randomly assigned conditions (combinations of carrier and nicotine concentrations).

CONDITION II: Participants attend up to 2 video or telephone conferences over 2 hours each with a minimum of 24 hours and maximum of 1 week between sessions. Participants take a fixed number of puffs on a nicotine-free condition and 3 randomly assigned conditions (combinations of carrier concentration and nicotine form).

ELIGIBILITY:
Inclusion Criteria:

* Current daily vapers of products containing nicotine
* No concurrent use of other tobacco products
* Self reported general good health
* No allergies - specifically known active untreated seasonal allergies that would interfere with smell or taste procedures
* No self-reported taste or smell deficits
* Not pregnant or lactating
* No medications known to interfere with taste/smell (i.e.: certain nasal sprays, nasal antihistamines, decongestants, antibiotics, medications containing zinc)
* Passing scores on the phenylthiocarbamine (PTC) and 6-n-propylthiouracil (PROP) smell and taste tests
* Access to video-conference or telephone
* Ability to store test products in a secure location away from children

Exclusion Criteria:

* Not current daily vapers
* Concurrent use of other tobacco products
* Self-reported fair or poor general health
* Allergies - active untreated seasonal allergies that would interfere with smell or taste procedures
* Self-reported taste or smell deficits
* Pregnant or lactating
* Medications known to interfere with taste/smell (i.e.: certain nasal sprays, nasal antihistamines, decongestants, antibiotics, medications containing zinc)
* Failing scores on the phenylthiocarbamine (PTC) and 6-n-propylthiouracil (PROP) smell and taste tests
* No access to video-conference or telephone
* Unable to store test products in a secure location away from children
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Adults unable to consent
* Adults unable to legally purchase tobacco products in New York (NY) state (18-20)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants from general population in the greater Buffalo area and are current daily vapers
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Sensory response measures | 2 years
  Will be assessed by product evaluation scale - Scale consists of 22 questions with #1 = Not at all - 7 = Extremely
Sensory response measure | 2 years
  gMLS rating of harshness, throat hit, and pleasantness.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J O'Connor, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States